CLINICAL TRIAL: NCT03625843
Title: Incorporation of Mindfulness Exercises to Reduce Anxiety and Pain During Urodynamic Testing: a Randomized Controlled Trial
Brief Title: Mindfulness Exercises to Reduce Anxiety and Pain During Urodynamic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Forrest Jellison, Principle Investigator, San Antonio Uniformed Services Health Education Consortium
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: c.2016.202d
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Stress Incontinence, Female; Overactive Bladder; Lower Urinary Tract Symptoms
Keywords: urodynamics
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfullness exercises (Experimental): Participate in mindfulness exercises prior to urodynamic studies (UDS). As a participant, you will be guided through a mindfulness meditation exercise by a licensed professional. During this exercise you will be asked to focus your attention on your breathing, physical sensations, and thoughts. This exercise will last for approximately 10 minutes.
  Interventions: Behavioral: Mindfulness exercises
- Control (No Intervention): Sitting quietly in a room alone.

INTERVENTIONS:
Behavioral: Mindfulness exercises
  Arms: Mindfullness exercises

SUMMARY:
In this pilot study the investigators attempt to answer the question, does mindfulness exercises before urodynamic testing reduce patient's perception of anxiety or pain?

DETAILED DESCRIPTION:
The subjects are being asked to consider participation in this research study. The purpose of this study is to see if incorporating mindfulness exercises prior to urodynamic studies (UDS) results in less pain, anxiety and discomfort.

The participants will be guided through a mindfulness meditation exercise by a licensed professional. During this exercise participants will be asked to focus attention on breathing, physical sensations, and thoughts. This exercise will last for approximately 10 minutes in which participants will not be asked to engage in any physical activity other than sitting and breathing. The participants will be randomly assigned to one of 2 treatment plans. Randomization is a process like flipping a coin and means the chance of being assigned to either of the plans. One treatment plan includes undergoing mindfulness exercises prior to your UDS evaluation. The other treatment plan includes simply undergoing the UDS evaluation.

After the participants UDS evaluation, questions will be asked about the urodynamic procedure. The participants will be asked to answer questions on a UDS and anxiety questionnaire which pertain to emotional and physical experiences during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urinary symptoms requiring urodynamic testing

  * Stress incontinence
  * Mixed incontinence
  * Urge incontinence
  * Overactive bladder
  * Urinary retention
  * Lower urinary tract symptoms
* Are Department of Defense (DoD) beneficiaries

Exclusion Criteria:

* Neurogenic bladder
* Interstitial cystitis
* Chronic bladder pain
* Inability to have urodynamics performed
* Are Not DoD beneficiaries
* Pregnant
* Lack capacity to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety during urodynamics as measured the STAI-6. | Day 1
  The STAI-6, State Trait Anxiety Inventory, is a validated questionnaire that measures anxiety. The total score from the STAI-6 will be used with a range of score from 4-24. Higher scores indicate higher level of anxiety.

SECONDARY OUTCOMES:
Positive and negative emotions as measured by the urodynamic questionnaire | Day 1
  The urodynamic questionnaire is clinically validated with participants self-reporting emotions fear, discomfort, embarrassment, and if the test was better or worse than expected. The questions are analyzed individually with score ranked on a likert scale of 1-4. Higher score indicate higher levels of that particular emotion.
Pain as measured by the VAS | Day 1
  The visual analog scale (VAS) for pain total score will be recorded. The minimum and Maximum scores range from 1-10. Higher scores indicate more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Forrest C Jellison, MD, Principal Investigator — San Antonio Uniformed Services Health Education Consortium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03625843/Prot_SAP_000.pdf